CLINICAL TRIAL: NCT04669457
Title: Prevention of Emergence Delirium in Pediatric Ambulatory Surgery: Single Blinded Randomized Control Study Comparing Intra-nasal Dexmedetomidine With Oral Midazolam.
Brief Title: Pediatric Delirium
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, R. Ian Richmond, Assistant Professor, Director of Clinical Operations, Dept of Anesthesiology and Perioperative Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H00021788
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Delirium
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The surgeon and post-operative nurses will be masked to the group allocation. Masking will only be revealed if medically necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intra-nasal Dexmedetomidine (Experimental): Subjects will receive Dexmedetomidine intra-nasally in the preoperative area. It will be administered at a dose of 1 mcg/kg, approximately 15-25 minutes before entering the operating room.
  Interventions: Drug: Intra-nasal Dexmedetomidine
- Oral Midazolam (Active Comparator): Subjects will receive Midazolam orally in the preoperative area. It will be administered at a dose of 0.5 mg/kg (with a maximum dose of 20 mg), approximately 10-15 minutes before entering the operating room.
  Interventions: Drug: Oral Midazolam

INTERVENTIONS:
Drug: Intra-nasal Dexmedetomidine — Subjects will receive Dexmedetomidine intra-nasally in the preoperative area. It will be administered at a dose of 1 mcg/kg, approximately 15-25 minutes before entering the operating room.
  Other Names: Precedex
  Arms: Intra-nasal Dexmedetomidine
Drug: Oral Midazolam — Subjects will receive Midazolam orally in the preoperative area. It will be administered at a dose of 0.5 mg/kg (with a maximum dose of 20 mg), approximately 10-15 minutes before entering the operating room.
  Other Names: Midazolam
  Arms: Oral Midazolam

SUMMARY:
Preventing emergent delirium in pediatric ambulatory surgery through preoperative use of intra-nasal Dexmedetomidine and oral Midazolam.

DETAILED DESCRIPTION:
Pediatric ambulatory patients will randomly be allocated to one of two groups. Group A which will receive Dexmedetomidine intra-nasally at a dose of 1 mcg/kg, approximately 15-25 minutes before entering the operating room or Group B which will receive Midazolam orally at a dose of 0.5 mg/kg (with a maximum dose of 20 mg), approximately 10-15 minutes before entering the operating room. Each subject will receive a Drug Acceptance scale, and Parental Separation Anxiety Scale (PSAS) mask Acceptance Scale to identify the differences in markers associated with pediatric delirium. End tidal Sevoflurane value during the surgery and at the time when patient leaves the OR, amount and dose of oral/rectal acetaminophen given in PACU, child's behavior for 48 hours post-operatively, and documented intake of oral analgesics will be collected to identify the reduced need for post-operative analgesia and behaviors associated with extended pediatric delirium.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 3 months to 9 years
* Scheduled to undergo a myringotomy
* American Society of Anesthesiologists (ASA) classification of I - II.

Exclusion Criteria:

* Subjects with unrepaired cardiac defects, including cyanotic congenital heart disease.
* Anyone age 10 years or older.
* Anyone with an ASA classification of III or higher.
* Non-English language speaker for whom short form consent is not available.

Ages: 3 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Time to onset of pediatric delirium | Zero minutes to 48 hours
  Time from when the patient is woken from anesthesia to the onset of delirium.
Time to offset of pediatric delirium | Zero minutes to 48 hours
  Time from onset of delirium to the offset of delirium.
Duration of pediatric delirium | Zero minutes to 48 hours
  Total time patient experiences delirium

SECONDARY OUTCOMES:
Drug Acceptance | 10-25 minutes prior to surgery
  The willingness of the subject to take the drug was assessed in the pre-operative area
Parental Separation Anxiety Scale (PSAS) | 0-48 hours
  Anxiety score was determined when the child was separated from the parents according to four levels.
Mask Acceptance Scale | 1-10 minutes prior to surgery
  The child's acceptance of the mask by the anesthesiologist was rated as follows.
End tidal Sevoflurane value | 0-12 hours
  During the surgery and at the time when patient leaves the OR End tidal Sevoflurane value will be documented.
Rescue analgesia in PACU | 0-6 hours post surgery
  The amount and dose of oral/rectal acetaminophen given in PACU was recorded.
Home Behavior Analysis | 12-48 hours
  The child's parents were given a diary to document their behavior for 48 hours post-operatively at home.
Oral analgesic use | Two days post-operative
  Document intake of oral analgesics like acetaminophen or ibuprofen

CONTACTS AND LOCATIONS:
Overall Officials: R. Ian Richmond, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared via publication as group data.